CLINICAL TRIAL: NCT05813327
Title: A Phase I/II Trial of Neoadjuvant ADI-PEG 20 in Combination With Ifosfamide and Radiotherapy in Soft Tissue Sarcoma (STS)
Brief Title: Neoadjuvant ADI-PEG 20 + Ifosfamide + Radiotherapy in Soft Tissue Sarcoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Polaris Group (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202305073
Record Dates: First submitted 2023-04-02; First posted 2023-04-14 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Soft Tissue Sarcoma; Sts; Sarcoma,Soft Tissue
Keywords: arginine starvation; ADI-PEG20; ifosfamide; radiotherapy; radiation therapy; ASS1 expression
MeSH Terms: conditions — Sarcoma; Ichthyosis, X-Linked | interventions — ADI PEG20; Ifosfamide; Radiotherapy; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Phase I: ADI-PEG 20 + ifosfamide + radiotherapy (Experimental): Patients will receive ADI-PEG 20 on Day -7 of Cycle 1 and Days 1, 8, and 15 of each of three 21-day cycles, and ifosfamide per dose escalation/de-escalation schedule on days 1 through 5 of each cycle. Mesna will be given on days 1 through 5 with ifosfamide as supportive care. Patients will also receive radiotherapy (XRT) starting on Week 4.
  Interventions: Drug: ADI PEG20; Drug: Ifosfamide; Radiation: Radiotherapy; Drug: Mesna
- Phase II: ADI-PEG 20 + ifosfamide + radiotherapy (Experimental): Patients will receive ADI-PEG 20 on Day -7 of Cycle 1 and Days 1, 8, and 15 of each of three 21-day cycles, and ifosfamide per the RP2D determined in Phase I of the study on days 1 through 5 of each cycle. Mesna will be given on days 1 through 5 with ifosfamide as supportive care. Patients will also receive radiotherapy (XRT) starting on Week 4.
  Interventions: Drug: ADI PEG20; Drug: Ifosfamide; Radiation: Radiotherapy; Drug: Mesna

INTERVENTIONS:
Drug: ADI PEG20 — ADI-PEG 20 will be given on an outpatient basis at a dose of 36 mg/m^2 via intramuscular injection into either the deltoid or gluteal muscle.
  Other Names: PEGylated arginine deiminase
Drug: Ifosfamide — Ifosfamide will be administered intravenously per package insert and institutional practice on Days 1 through 5 of all 3 cycles.
  Other Names: ifex
Radiation: Radiotherapy — Radiotherapy will begin on C2D1 and will continue as per institutional practice.
Drug: Mesna — Mesna will be administered for supportive care either intravenously or by mouth per package insert and institutional practice on Days 1 through 5 of all 3 cycles.
  Other Names: sodium 2-mercaptoethane sulfonate

SUMMARY:
In this study, patients with soft tissue sarcoma (STS) will receive ADI-PEG 20 and ifosfamide in combination with radiation as neoadjuvant therapy. In phase I of the study, up to 5 dose levels will be tested to find the recommended phase II dose (RP2D), after which patients enrolling to phase II will be treated at that dose level to assess efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically proven diagnosis of grade 2-3 (intermediate or high grade) soft tissue sarcoma of the trunk or extremities with size ≥5 cm by clinical or radiographic assessment that is appropriate for ifosfamide therapy. Patients must be planning to undergo treatment with curative intent.
* Patients with sufficient tumor tissue for correlative analyses. Patients without sufficient tissue may be allowed to enroll on a case-by-case basis with permission of sponsor-investigator.
* Staging workup shows no definitive evidence of distant metastasis and there is planned definitive surgical resection of the primary tumor.
* At least 18 years of age at time of consent.
* ECOG performance status ≤ 1
* Adequate bone marrow, coagulation, and organ function as defined below:

  * Absolute neutrophil count ≥ 1.5 K/cumm
  * Platelets ≥ 100 K/cumm
  * Hemoglobin ≥ 9 g/dL (no transfusions within 7 days of C1D-7)
  * International Normalized Ratio (INR) ≤ 1.5 x IULN or prothrombin time (PT) ≤ 1.5 x IULN, and partial thromboplastin time (aPTT or PTT) ≤ 1.5 x IULN (inclusion only applicable to subjects not using anticoagulation).
  * Total bilirubin ≤ 1.5 x IULN (except for patients with Gilbert's Syndrome, who must have a total bilirubin <3 mg/dL)
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN
  * Creatinine clearance ≥ 60 mL/min/1.73^2 by MDRD
* The effects of the study therapy on the developing human fetus are unknown. For this reason and because chemotherapeutics are known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and 12 months after completion of the study. Should a woman or female partner become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Highly effective methods of birth control are defined as those that results in a low failure rate (that is, <1% per year) when used consistently and correctly, such as implants, injectables, combined oral contraceptives, some intrauterine contraceptive devices (IUDs), partner or a vasectomized partner. Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study intervention. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant. Exceptions: Exceptions: Females not of child-bearing potential due to surgical sterilization (at least 6 weeks following tubal ligation, hysterectomy, or surgical bilateral oophorectomy with or without hysterectomy) confirmed by medical history; or postmenopausal female. A postmenopausal female is a female meeting either of the following criteria: Spontaneous amenorrhea for at least 12 months, not induced by a medical condition such as anorexia nervosa and not taking medications during the amenorrhea that induced the amenorrhea (for example, oral contraceptives, hormones, gonadotropin releasing hormone, antiestrogens, selective estrogen receptor modulators [SERMs], or chemotherapy). Spontaneous amenorrhea for 6 to 12 months and a follicle-stimulating hormone (FSH) level >40 IUnits/L
* Ability to understand and willingness to sign an IRB approved written informed consent document.

Exclusion Criteria:

* Pure well-differentiated liposarcoma, low grade STS, Kaposi sarcoma, bone sarcomas, cartilage sarcomas, or GIST.
* Definitive clinical or radiologic evidence of metastatic disease; indeterminate lung nodules less than 5 mm are acceptable.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Currently receiving any other investigational agents.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to ADI-PEG 20, ifosfamide, PEGylated compounds, or other agents used in the study.
* Prior systemic chemotherapy for the study cancer (sarcoma); note that prior chemotherapy for a different cancer (including a different sarcoma) is allowable if given greater than three years prior. However, unresolved toxicities from prior anti-tumor therapy, defined as not having resolved to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grade 0 or 1, or to levels dictated in the eligibility criteria with the exception of alopecia (Grade 2 or 3 toxicities from prior antitumor therapy that are considered irreversible [defined as having been present and stable for > 6 months] may be allowed if they are not otherwise described in the exclusion criteria AND there is agreement to allow by the sponsor-investigator.
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields.
* Clinically significant bleeding within 4 weeks of C1D-7, current use of direct thrombin inhibitors unless these medications can be safely discontinued 14 days prior to C1D-7. Note: Low molecular weight heparin and factor Xa inhibitors are permitted.
* Concomitant use of the below medications is restricted during the study:

  * All herbal medicines (e.g., St. John's wort), and supplements, within the 6 days prior to C1D-7. Standard adult multi-vitamin is allowed.
  * CYP2C8 substrates with a narrow therapeutic window within the 6 days prior to C1D-7.
  * No live vaccines within 6 days of C1D-7.
* Patients with active infection requiring IV antibiotics within 2 weeks of C1D-7
* The patient has a serious cardiac condition, such as congestive heart failure; New York Heart Association Class III/IV heart disease; unstable angina pectoris, cardiac stenting within 6 months of C1D-7; myocardial infarction within 6 months of C1D-7; valvulopathy that is severe, moderate, and deemed clinically significant; or arrhythmias that are symptomatic or require treatment.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum pregnancy test within 7 days of C1D-7.
* Patients with known active Hepatitis B or C or HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-03-14 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
Treatment-related serious adverse event (SAE) rate | From start of study treatment through 30 days from end of neoadjuvant treatment (estimated to be 14 weeks)
  An adverse event is considered serious if, in the view of the investigator, it results in any of the following:
  * Death
  * A life threatening adverse event
  * Inpatient hospitalization or prolongation of existing hospitalization
  * A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
  * A congenital anomaly/birth defect
  * Any other important medical event that does not fit the criteria above but, based upon appropriate medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed above
Recommended Phase II dose (Phase I only) | From start of study treatment through 2 cycles of treatment (estimated to be 7 weeks)
  The MTD is defined as the highest dose level at which no more than 1 out of 6 patients experienced DLT at the end of Cycle 2. Dose escalations will proceed until the MTD has been reached or until Dose Level 3, and this dose level will then be defined as the Recommended Phase 2 Dose (RP2D).

SECONDARY OUTCOMES:
Percent necrosis in final surgical specimen | At time of surgical resection (estimated to be 16 weeks)
  Defined as the proportion of patients with a necrosis in the final surgical specimen.
Pathologic complete response (pCR) in final surgical specimen | At time of surgical resection (estimated to be 16 weeks)
  Defined as the proportion of patients with a pCR confirmed in the final surgical specimen.
Percent local failure (%LF) | At 2 years from surgical resection (estimated to be 120 weeks)
  Defined as the proportion of patients with a local failure, which is either local tumor recurrence or local tumor progression.
Disease free survival (DFS) | At 2 years from surgical resection (estimated to be 120 weeks)
  Defined as the time from start of treatment to time of recurrence or death, whichever occurs first.
Overall survival (OS) | At 2 years from surgical resection (estimated to be 120 weeks)
  Defined as the time from start of treatment to death from any cause.
Response rate per RECIST 1.1 | After completion of treatment but prior to surgery (estimated to be 10 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Mia Weiss, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu